CLINICAL TRIAL: NCT00418613
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study, Conducted Under In-House Blinding Conditions of MK0633 in Patients With COPD
Brief Title: A Research Study of MK0633 in Patients With Chronic Obstructive Pulmonary Disease (COPD)(0633-009)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0633-009; MK0633-009; 2006_509
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): MK0633
  Interventions: Drug: MK633
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo (unspecified)

INTERVENTIONS:
Drug: MK633 — MK0633 100mg capsules qd for a 12-wk treatment period.
  Arms: 1
Drug: Comparator: Placebo (unspecified) — MK0633 100mg Pbo capsules for a 12-wk treatment period
  Arms: 2

SUMMARY:
A clinical study to evaluate the efficacy and safety of MK0633 in patients with Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Documented COPD defined by clinical history and spirometry, with symptoms including dyspnea, wheezing, chest tightness, cough, sputum production, or nocturnal awakening
* Male or postmenopausal females 40 -75 years of age

Exclusion Criteria:

* Impaired renal function
* History of chronic liver disease or persistent liver function test (LFT) abnormalities
* History of recent cardiovascular clinical event
* Evidence of another clinically significant, active pulmonary disorder such as bronchiectasis or asthma

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pulmonary function test data | Measured over 12 weeks

SECONDARY OUTCOMES:
Overall daytime symptoms score, total daily beta agonist use, and Chronic Respiratory Disease Questionnaire (CRQ) score | Measured over 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Bernstein JA, Liu N, Knorr BA, Smugar SS, Hanley WD, Reiss TF, Greenberg S. MK-0633, a potent 5-lipoxygenase inhibitor, in chronic obstructive pulmonary disease. Respir Med. 2011 Mar;105(3):392-401. doi: 10.1016/j.rmed.2010.09.021. Epub 2010 Nov 13. PMID 20970976